CLINICAL TRIAL: NCT05716230
Title: Bowel Function and Associated Risk Factors for Bowel Dysfunciton in Preschool and Early Childhood in Patients With Anorectal Malformation
Brief Title: Bowel Function and Associated Risk Factors for Bowel Dysfunciton in Patients With Anorectal Malformation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Weibing Tang, Director, Nanjing Children's Hospital
Other Study IDs: NanjingCH0109
Record Dates: First submitted 2023-01-09; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Bowel Dysfunction
Keywords: anorectal malformation; Bowel function; risk factors
MeSH Terms: conditions — Intestinal Diseases; Anorectal Malformations

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: bowel function score questionnaire survey — Bowel function score(BFS, total 20 points) was approved by Rintala in 1995, and patients with a score ≥ 17 were considered to have normal bowel habits. 7 items were in BFS, including the ability to hold back defecation, feeling/reporting the urge to defecate, frequency of defecation, soiling, accidents, constipation. In December 2022, BFS questionnaire surveys were conducted on children with ARM who underwent surgical repair between January 2017 and December 2019 at Children's Hospital of Nanjing Medical University.

SUMMARY:
The present study was designed to evaluate bowel function in preschool and early childhood in a large number of patients with anorectal Malformation and to identify the associated risk factors for bowel dysfunction.

DETAILED DESCRIPTION:
Anorectal malformation (ARM) is a type of congenital malformation resulting from post-embryonic intestinal dysgenesis, occurring in about 1 in 5000 cases.Surgery is an effective means of treating ARM,which includes reconstruction of the anus and treatment of associated deformities. However, even with reconstruction of the anus, most children still have serious complications, such as constipation, fecal incontinence, urinary incontinence, and sexual dysfunction, in the mid-to-long postoperative period.A lot of studies have been designed to explore the trend toward normal bowel habits from preschool and early childhood age to adolescence or adult; however, no apparent improvement in bowel habits was completely confirmed. In contrast, many reports have shown that poor bowel function in preschool and early childhood may lead to social problems and depression in adolescence and adult.The reasons for bowel dysfunction of ARM in preschool and early childhood were complicated and undefined,including associated malformations, the type of ARM, and the development of the perianal sphincter,etc.The bowel function score (BFS) is currently used to assess mid- and long-term anal function in patients with ARM, and comprises seven major categories (e.g., self-perception, fecal control, stool collection, and social problems) with a total of 20 points, or less than 17 points, for the presence of anal weakness (11-17 points, for the general weakness, or less than 11 points, for the severe weakness) .Therefore,bowel function at preschool and early childhood should be evaluated in a large number of patients with ARM and the associated risk factors for bowel dysfunction should also be assessed. The present study was designed to evaluate bowel function in preschool and early childhood in a large number of patients with ARM and to identify the associated risk factors for bowel dysfunction using BFS.

ELIGIBILITY:
Inclusion Criteria:

Anorectal malformation >4 years old

Exclusion Criteria:

Down syndrome patients <4 years

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ARM who were performed with surgery.The follow-up age was more than 4 years old.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-01-29 (Actual); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
bowel function score in partipants with ARM | through study completion, an average of 6 year
  approved by Rintala in 1995, and patients with a score ≥ 17 were considered to have normal bowel habits

SECONDARY OUTCOMES:
Sacral ratio in partipants with ARM | through study completion, an average of 6 year
  test by X ray

OTHER OUTCOMES:
Number of partipants with every type of ARM | through study completion, an average of 6 year
  confirmed in surgery
age at surgery of partipants with ARM | through study completion, an average of 6 year
  age at surger
Number of partipants performed with every surgical method | through study completion, an average of 6 year
  Posterior sagittal approach to anoplasty or Anterior sagittal approach to anoplasty or Laparoscopic assisted anoplasty
Number of partipants with abnormal spinal cord | through study completion, an average of 6 year
  tethered cord or other
Number of partipants with reoperation | through study completion, an average of 6 year
  re-anoplasty

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Tang, Dr, Study Director — Children's Hospital of Nanjing Medical University
Locations (1):
- Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Lu C, Pan S, Chen H, Tang W. Bowel function and features of bowel dysfunction in preschool children with anorectal malformation type rectoperineal and rectovestibular fistula. Eur J Pediatr. 2024 Feb;183(2):599-610. doi: 10.1007/s00431-023-05306-4. Epub 2023 Nov 8. PMID 37935997